CLINICAL TRIAL: NCT05327374
Title: Diagnosis of Acute Heart Failure in Chronic Obstructive Pulmonary Disease Exacerbation Using the Inferior Vena Cava Collapsibilty Index
Brief Title: Use of ΔIVC for Early Diagnosis of AHF in AECOPD
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Other Study IDs: ΔIVC /AHF/ AECOPD
Record Dates: First submitted 2022-03-14; First posted 2022-04-14 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Acute Decompensated Heart Failure; COPD Exacerbation
Keywords: COPD; Acute Heart Failure; Inferior vena cava; Ultrasound; Collapsibility index
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AHF-group: patients with AECOPD and acute heart failure
  Interventions: Diagnostic Test: calculation of the inferior vena cava collapsibility index
- non AHF-group: patients with AECOPD without acute heart failure
  Interventions: Diagnostic Test: calculation of the inferior vena cava collapsibility index

INTERVENTIONS:
Diagnostic Test: calculation of the inferior vena cava collapsibility index — the ΔIVC was calculated by the emergency physician who was blinded from the patient's medical history using the formula ((IVCmax-IVCmin)/IVCmax) X100.A cutoff of 15% was used to define the presence(<15%) or absence(>15%) of heart failure

SUMMARY:
Acute Heart failure (AHF) is a common cause of acute exacerbation of chronic obstructive pulmonary disease (AECOPD).

This association is frequently underestimated with regard to the difficulty of clinical diagnosis.

The investigators expect that the application of the inferior vena cava collapsibility index (ΔIVC)could be useful in this issue.

DETAILED DESCRIPTION:
Acute heart failure (AHF) is a common cause of COPD exacerbation however its role is very often underestimated. Until now, the use of echocardiography and some invasive hemodynamic exploration techniques such as the Swanganz catheter has been stated as reference. Other noninvasive diagnostic methods have been studied, such as systolic time intervals and Valsalva maneuver, but their application still difficult in patients with COPD exacerbation, especially in emergency department (ED) settings. the study aimed to evaluate the performance of a new diagnostic technique based on the measurement of the ΔIVC for the early identification of AHF in patients presenting to the ED with acute COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* patient with history of COPD and admitted to the emergency departement for AECOPD

Exclusion Criteria:

* impossibility to give consent to participate in the study, non consent patients
* post traumatic dyspnea
* instable hemodynamic or neurological status

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with history of COPD admitted to the emergency departmet for AECOPD and stable hemodynamic status
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
the performance of ΔIVC in the diagnosis of acute heart failure | 1 day
  the accuracy of ΔIVC in the diagnosis of heart failure measured by sensitivity ,specificity, and area under the roc curve

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — University of Monastir
Locations (3):
- Tunisia (3):
  - CHU Fattouma Bourguiba, Monastir
  - Emergency Departement, Monastir
  - Emergency department of fattouma bourguiba university hospital, Monastir

IPD SHARING:
Plan to Share IPD: Undecided